CLINICAL TRIAL: NCT05278676
Title: A Single and Multiple Dose Pharmacokinetic Study of Dotinurad in Chinese Healthy Subjects
Brief Title: A Single and Multiple Dose Study of Dotinurad in Chinese Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FYU-981-J086-001
Record Dates: First submitted 2022-02-18; First posted 2022-03-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — dotinurad

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A Single Dose: Dotinurad (Experimental): Participants will receive dotinurad 1 milligram (mg) (1*1 mg tablet) as a single oral dose after 10-hour fasting on Day 1 in the morning.
  Interventions: Drug: Dotinurad
- Cohort B Multiple Dose: Dotinurad (Experimental): Participants will receive dotinurad 4 mg (2*2 mg tablets) as a single oral dose after 10-hour fasting on Day 1 in the morning. A washout period of 3 days will be maintained after single dose on Day 1 and then participants will receive dotinurad 4 mg (2*2 mg tablets) after 10-hour fasting from Day 4 to Day 10 once daily in the morning.
  Interventions: Drug: Dotinurad
- Cohort C Single Dose: Dotinurad (Experimental): Participants will receive dotinurad 10 mg (5*2 mg tablets) as a single oral dose after 10-hour fasting on Day 1 in the morning.
  Interventions: Drug: Dotinurad

INTERVENTIONS:
Drug: Dotinurad — Dotinurad oral tablet.
  Other Names: FYU-981

SUMMARY:
The primary purpose of this study is to evaluate the pharmacokinetics (PK) of dotinurad following single and multiple oral doses of dotinurad in Chinese healthy male and female participants.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy Chinese participants living in China.
2. Non-smoking, male or female, age greater than or equal to (>=) 18 years and less than or equal to (<=) 45 years old at the time of informed consent.
3. Participants with serum uric acid level less than >=5.5 milligrams per decilitre (mg/dL) at Screening (Cohort B only).

Key Exclusion Criteria:

1. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [β-hCG] or human chorionic gonadotropin [hCG] test). A separate baseline assessment of serum β-hCG (or hCG) or urine pregnancy test is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
2. Females of childbearing potential.
3. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing.
4. Evidence of disease that may influence the outcome of the study within 4 weeks before dosing; example, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism.
5. Any history of gastrointestinal surgery that may affect PK profiles of dotinurad, example, hepatectomy, nephrectomy, digestive organ resection at Screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Single-dose Part, Cmax: Maximum Observed Concentration for Dotinurad | Day 1: 0-48 hours post dose
Single-dose Part, Tmax: Time at Which the Highest Drug Concentration Occurs for Dotinurad | Day 1: 0-48 hours post dose
Single-dose Part, t1/2: Terminal Elimination Phase Half-life for Dotinurad | Day 1: 0-48 hours post dose
Single-dose Part, AUC0-t: Area Under the Concentration-time Curve From Zero Time to Time of Last Quantifiable Concentration for Dotinurad | Day 1: 0-48 hours post dose
Single-dose Part, AUC0-24h: Area Under the Concentration-time Curve From Zero Time to 24 hours for Dotinurad | Day 1: 0-24 hours post dose
Single-dose Part, AUC0-inf: Area Under the Concentration-time Curve From Zero Time Extrapolated to Infinite Time for Dotinurad | Day 1: 0-48 hours post dose
Single-dose Part, CL/F: Apparent Total Clearance Following Oral Administration for Dotinurad | Day 1: 0-48 hours post dose
Single-dose Part, Vz/F: Apparent Volume of Distribution at Terminal Phase for Dotinurad | Day 1: 0-48 hours post dose
Single-dose Part, kel: Elimination Rate Constant for Dotinurad | Day 1: 0-48 hours post dose
Single-dose Part, MRT0-t: Mean Residence Time From Zero Time to Time of Last Quantifiable Concentration on Single Dose for Dotinurad | Day 1: 0-48 hours post dose
Multiple-dose Part, Css,max: Maximum Observed Concentration at Steady State for Dotinurad | Day 10: 0-72 hours post dose
Multiple-dose Part, Css,min: Minimum Observed Concentration at Steady State for Dotinurad | Day 10: 0-72 hours post dose
Multiple-dose Part, Css,av: Average Steady-state Concentration for Dotinurad | Day 10: 0-72 hours post dose
Multiple-dose Part, tss,max: Time at Which the Highest Drug Concentration Occurs at Steady State for Dotinurad | Day 10: 0-72 hours post dose
Multiple-dose Part, t1/2: Terminal Elimination Phase Half-life for Dotinurad | Day 10: 0-72 hours post dose
Multiple-dose Part, AUC0-τ: Area Under the Concentration-time Curve Over the Dosing Interval on Multiple Dosing for Dotinurad | Day 10: 0-72 hours post dose
Multiple-dose Part, CLss/F: Apparent Total Clearance Following Oral Administration at Steady State for Dotinurad | Day 10: 0-72 hours post dose
Multiple-dose Part, Vz/F: Apparent Volume of Distribution at Terminal Phase for Dotinurad | Day 10: 0-72 hours post dose
Multiple-dose Part, kel: Elimination Rate Constant for Dotinurad | Day 10: 0-72 hours post dose
Multiple-dose Part, MRT: Mean Residence Time for Dotinurad | Day 10: 0-72 hours post dose
Multiple-dose Part, Rac(AUC0-24h): Accumulation Ratio for AUC(0-24h) | Day 10: 0-24 hours post dose
Multiple-dose Part, Rac(Cmax): Accumulation Ratio for Cmax | Day 10: 0-72 hours post dose
Multiple-dose Part, PTF: Peak-trough Fluctuation | Day 10: 0-72 hours post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui District Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Liu Y, Chen Q, Sun H, Cai C, Kawamura K, Kokan R, Nomoto M. A Single- and Multiple-Dose Study to Characterize the Pharmacokinetics and Safety of Dotinurad in Healthy Chinese Adults. Clin Drug Investig. 2025 Dec;45(12):957-966. doi: 10.1007/s40261-025-01496-x. Epub 2025 Oct 19. PMID 41111126